CLINICAL TRIAL: NCT02143167
Title: RETRAP - A Double Blind, Randomized, Placebo Controlled Study of the Effect of the Combination of Resistance Training and Prolonged Release Fampridine in Patients With Multiple Sclerosis
Brief Title: Resistance Training and Amino Pyridine in Multiple Sclerosis
Acronym: RETRAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other); Biogen (Industry)
Responsible Party: Principal Investigator, Henrik Boye Jensen, Medical doctor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RETRAP; 2011-002959-34 (EudraCT Number)
Record Dates: First submitted 2014-05-09; First posted 2014-05-20 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SR-fampridine/placebo (Experimental): 24 weeks of SR-fampridine followed by four weeks of inactive placebo.
  Interventions: Drug: SR-fampridine; Drug: Placebo
- Placebo/SR-fampridine (Experimental): 24 weeks of inactive placebo followed by four weeks of SR-fampridine
  Interventions: Drug: SR-fampridine; Drug: Placebo

INTERVENTIONS:
Drug: SR-fampridine — One arm receives SR-fampridine 10 mg BID for 24 weeks followed by four weeks of inactive placebo BID.
  The other arm receives placebo BID for 24 weeks followed by four weeks of SR-fampridine 10 mg BID for four weeks.
  Other Names: Fampyra
Drug: Placebo

SUMMARY:
Prolonged-release fampridine (SR-fampridine) can improving walking capacity in approximately 40% of MS patients suffering from this by overcoming partly or total conduction block due to demyelination.

Resistance training has been shown to provide the same kind of benefits for patients by targeting the muscular component of the motor unit. Thus by combining the two it is likely to see an synergistic effect.

This trial is designed as a double blind, randomized placebo controlled trial with subsequent cross-over.

Participants in the two arms will go through the same progressive training program targets at the lower limbs. For 24 weeks one group receives SR-fampridine and the other receives placebo. in the the end there is another four weeks of training after cross-over has been performed.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsing remitting multiple sclerosis (RRMS), secondary progressive multiple sclerosis (SPMS) or primary progressive multiple sclerosis (PPMS) fulfilling the McDonald criteria
* Expandend Disability Status Scale (EDSS) 3-6.5
* Pyramidal Functional Score ≥ 2
* Participants must be able to transport self to gym and to the University of Southern Denmark
* Participants must be able to complete T25FW and SSST
* Fertile female participants are obliged to use hormonal contraceptive measures

Exclusion Criteria:

* History of epileptic seizures
* MS relapse or change in disease modifying treatment (DMT) within 60 days
* Cancer within five years
* Blood pressure ≥ 160/100
* Severe arrhythmia or ischaemic heart disease or unexplained abnormal cardiac auscultation
* ≥ ALT 90 U/l, ≥ BSP 210 U/l, ≥ γ-GT 230 U/l
* GFR < 80 ml/min.
* History of severe pulmonary disease or unexplained abnormal pulmonary auscultation
* Pregnancy
* Breastfeeding
* Allergy to substances contained in prolonged release Fampridine tablets
* Concomitant treatment with carvedilol, propranolol or metformin.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Muscle power in the lower limbs | Muscle power will be measured after 14 weeks of resistance training.
  Muscle power in the lower limbs is measured by dynamometry pre and post resistance training

SECONDARY OUTCOMES:
Activity | Accelerometry is measured after 14 weeks of resistance training
  Activity measured by accelerometry.
Walking capacity | Walking capacity is measured after 26 weeks of resistance training
  Walking capacity measured by the Six Spot Step Test (SSST)
Walking speed | Walking speed is measured after 26 weeks of resistance training
  Walking speed measured by the Timed 25 Foot Walk (T25FW) and the 6-Minute Walking Test (6MWT)
Functional capacity in the lower limbs | Funcyional capacity in the lower limbs is measured after 26 weeks of resistance training
  Functional capacity measured by the Chair Stand Test (CST)
Self rated walking capacity | Self rated walking capacity is measured after 26 weeks of resistance training
  Self rated walking capacity measured by the 12-Item Multiple Sclerosis Walking Scale (MSWS12)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik B Jensen, MD, Principal Investigator — University of Southern Denmark
Locations (4):
- Denmark (4):
  - Sydvestjysk Sygehus, Esbjerg
  - Odense University Hospital, Odense
  - Sygehus Sønderjylland, Sønderborg
  - Sygehus Lillebælt, Vejle

REFERENCES:
- [Background] Dalgas U, Stenager E, Jakobsen J, Petersen T, Hansen HJ, Knudsen C, Overgaard K, Ingemann-Hansen T. Resistance training improves muscle strength and functional capacity in multiple sclerosis. Neurology. 2009 Nov 3;73(18):1478-84. doi: 10.1212/WNL.0b013e3181bf98b4. PMID 19884575
- [Background] Goodman AD, Brown TR, Edwards KR, Krupp LB, Schapiro RT, Cohen R, Marinucci LN, Blight AR; MSF204 Investigators. A phase 3 trial of extended release oral dalfampridine in multiple sclerosis. Ann Neurol. 2010 Oct;68(4):494-502. doi: 10.1002/ana.22240. PMID 20976768
- [Background] Goodman AD, Brown TR, Krupp LB, Schapiro RT, Schwid SR, Cohen R, Marinucci LN, Blight AR; Fampridine MS-F203 Investigators. Sustained-release oral fampridine in multiple sclerosis: a randomised, double-blind, controlled trial. Lancet. 2009 Feb 28;373(9665):732-8. doi: 10.1016/S0140-6736(09)60442-6. PMID 19249634